CLINICAL TRIAL: NCT00005997
Title: Phase II and Pharmacokinetic Trial of Rebeccamycin Analog in Hepatobiliary Cancers
Brief Title: Rebeccamycin Analogue in Treating Patients With Advanced Liver and/or Biliary Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual for Cohort II
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Afshin Dowlati MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWRU2299; U01CA063200 (NIH); P30CA043703 (NIH); CWRU-2299 (Other: Case Comprehensive Cancer Center); NCI-96
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer
Keywords: localized unresectable adult primary liver cancer; advanced adult primary liver cancer; unresectable gallbladder cancer; unresectable extrahepatic bile duct cancer; adult primary hepatocellular carcinoma; cholangiocarcinoma of the gallbladder; cholangiocarcinoma of the extrahepatic bile duct; adult primary cholangiocellular carcinoma
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — becatecarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: becatecarin — Cohorts of 3-6 patients receive escalating doses of rebeccamycin analogue until the maximum tolerated dose (MTD) is determined.
  Other Names: DEAE-rebeccamycin; rebeccamycin analogue; rebeccamycin analogue, tartrate salt

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of rebeccamycin analogue in treating patients who have advanced liver and/or biliary cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with advanced hepatobiliary carcinoma treated with rebeccamycin analogue.
* Assess the toxicity associated with this drug in this patient population.
* Evaluate the survival of this patient population treated with this drug.
* Determine the pharmacokinetics of this drug in this patient population.

OUTLINE: This is a partial dose-escalation study.

Patients receive rebeccamycin analogue IV over 1 hour daily on days 1-5. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are assigned to 1 of 2 cohorts according to hepatic dysfunction. (Cohort I closed to accrual as of 11/1/03.)

* Cohort I (closed to accrual as of 11/1/03): Patients receive a fixed dose of rebeccamycin analogue.
* Cohort II: Cohorts of 3-6 patients receive escalating doses of rebeccamycin analogue until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 6-37 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced hepatobiliary carcinoma not amenable to conventional surgery

  * Gall bladder carcinoma
  * Cholangiocarcinoma
  * Carcinoma of the ampulla
  * Hepatocellular carcinoma (eligible for cohort II only)
* Measurable disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Bilirubin less than 3 mg/dL

  * Cohort I (closed to accrual as of 11/1/03)

    * Bilirubin no greater than 1.5 mg/dL
    * AST no greater than 2.5 times upper limit of normal (ULN)
  * Cohort II

    * Bilirubin greater than 1.5 mg/dL and less than 3 mg/dL OR
    * Bilirubin no greater 1.5 mg/dL AND AST greater than 2.5 times ULN

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for cholangiocarcinoma or hepatobiliary carcinoma

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent combination antiviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 1999-04; Primary Completion 2005-04 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Determine the response rate in patients with advanced hepatobiliary carcinoma treated with rebeccamycin analogue. | Patients are followed every 3 months.

SECONDARY OUTCOMES:
Assess the toxicity associated with this drug in this patient population. | Patients are followed every 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Dowlati A, Posey J, Ramanathan RK, Rath L, Fu P, Chak A, Krishnamurthi S, Brell J, Ingalls S, Hoppel CL, Ivy P, Remick SC. Phase II and pharmacokinetic trial of rebeccamycin analog in advanced biliary cancers. Cancer Chemother Pharmacol. 2009 Dec;65(1):73-8. doi: 10.1007/s00280-009-1005-x. Epub 2009 Apr 28. PMID 19399502
- [Result] Dowlati A, Posey J, Ramanathan RK, et al.: Multicenter phase II and pharmacokinetic study of rebeccamycin analogue (RA) in advanced biliary cancers. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1070, 2003.